CLINICAL TRIAL: NCT02077101
Title: Representations and Acceptability of HIV Therapeutic Vaccine in a Cohort of HIV-1 Infected Outpatients Followed at Hospital : Multicentric Interventional Study Qualitative and Quantitative
Brief Title: Representations and Acceptability of HIV Therapeutic Vaccine in a Cohort of HIV-1 Infected Outpatients Followed at Hospital
Acronym: RAVVIH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Collaborators: Saint-Louis Hospital, Paris, France (Other); INSERM UMR912-SE4S, Marseille, France (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 2013/35
Record Dates: First submitted 2014-02-21; First posted 2014-03-04 (Estimated); Last update posted 2015-01-19 (Estimated); Status verified 2015-01

CONDITIONS: HIV
Keywords: HIV; Therapeutic vaccine; acceptability; representations
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quantitative study group (Other): Patients complete questionnaires validated and published in the literature: Brief IPQ R and HIV PROQOL [28, 29]. The questionnaire RAVVIH therapeutic vaccine has been designed from the literature review and advice of the Scientific Council in particular Dr. Pierre Verger social scientist vaccination and experts on the perception of patients. It was tested on a sample of 15 PWLHA
  Interventions: Other: Questionnaire
- Qualitative study group (Other): An interview guide was developed from the literature and expert community. Data will be collected through qualitative interviews with a psychologist trained to conduct interviews. Volunteers will be recruited according to the different categories of people representative of the HIV population in France.
  These interviews will be conducted at the Foch Hospital. The physician investigator propose participation in the investigation and agree on a day appointment with the psychologist. Consent will be collected at that time after reading the prospectus . All interviews will be recorded orally with the agreement of the participants , and transcribed in full . They will be completely anonymous .
  The average length of the interviews will be 45-60 minutes. Textual data from these interviews will be analysis.
  Interventions: Other: Interview

INTERVENTIONS:
Other: Questionnaire
  Arms: Quantitative study group
Other: Interview
  Arms: Qualitative study group

SUMMARY:
The main objective of the study is to assess the acceptability of a future therapeutic vaccine against HIV in patients living with HIV-1.

Secondary objectives concern the validation of a specific questionnaire for self-perception and acceptability of therapeutic vaccination against HIV-1 (RAVVIH), the development of a composite score for acceptability based on this questionnaire, and the analysis of critical factors related to: representations of vaccination in general, representations of therapeutic vaccination specific to HIV, perception of disease severity, health-related quality of life, doctor-patient relationship.

DETAILED DESCRIPTION:
Since 2000, the study of the acceptability of HIV vaccine candidates is one of four major areas recommended by the WHO. Presently, there are several studies in HIV field on the theme " Cure ". However, no study has yet addressed the question of the acceptability of therapeutic vaccine candidates against HIV who are currently already in clinical trials phase 2 and 3 In addition, many aspects of the disease, its treatment and living conditions of PLWHA could affect the acceptability of such a vaccine

Description of the study population :

The study population has the characteristics of the HIV population living in France [ 26, 27 ] .The French population reported by the database of the French Hospital in 2011 FHDH comparable to the population of their study ( three centers combined ) :- 36% of MSM- 9.1% of injection drug users (IDUs) 45% of heterosexuals : Europe including France 23.7% of immigrants from sub-Saharan Africa. 88 % were receiving antiretroviral therapy and 95% are undetectable .- 40 % are between 40-49 years

Description of the research methodology

Quantitative study : Patients complete questionnaires validated and published in the literature: Brief IPQ R and HIV PROQOL[ 28, 29 ] .The questionnaire RAVVIH therapeutic vaccine has been designed from the literature review , and the opinions ofScientific Council in particular Dr. Pierre Verger social scientist vaccination and experts on the perception of patients. It was tested on a sample of 15 PHAs.The questionnaire takes into account several important dimensions that could affect therapeutic vaccine acceptability :

1. the individual history , ARV treatment (tolerance ) and the perception of related adverse symptoms treatment
2. compliance with respect to ARV treatment
3. the quality of the relationship of the person with his or her physician ( referent , general ) and the level ofit gives them confidence ; 4 ) the level of social support person (unlike its isolation ) that may explain the desire to participate in a trial (more attention in the context of a trial , for example ... ) 5 ) managing the secret of his illness ( to avoid taking daily treatment with a vaccine therapy, can be a way to reduce the opportunities to reveal his illness ... )6) the perception of the seriousness of his illness.T

Qualitative study : A group of 20 patients will be offered a qualitative interview with a psychologist. The interview guide was developed from the literature and expert community. Volunteers will be recruited according to the different categories of people representative of the HIV population in France.

Study participation is approximately 30 minutes, including the presentation of protocol and the charging time of the questionnaire.

After giving consent in the study, the patient may at any time withdraw it and end its participation.

Paper questionnaires completed by the patients will be considered as source documents for this study and the patient's medical record where the following data will be collected (date of birth, viral load , therapy; vaccination status , mode of infection , nadir CD4 ,CD4 count , year of diagnosis , year of start of HAART, HBV and HCV co-infection status).

Quality assurance plan / Study Monitoring and Auditing :

This study will follow the monitoring and auditing guidelines designed by the sponsor in order to ensure agreement with good clinical practices recommendations.

Study monitoring and source data verification :

Monitoring will be achieved by a representative from the sponsor (Clinical Research Delegate) who will perform on-site visits during which s/he will compare data from the observation booklet with source data in order to assess its completeness. The clinical research delegate will ensure that, via frequent communication (either by mail, phone, fax, and email), the research is in agreement with the protocol and complies with regulation.

The site closing visit will be performed by the Clinical Research Delegate.

Site Monitoring : The national regulatory board and/or the representatives of the sponsor's Clinical Quality Board will be able to request access to source data, observation booklets, and all study documentation during site auditing or inspection. The investigator has to guarantee unhindered direct access to all the above-mentioned documentation and collaborate fully to site auditing and inspections. Medical files and all study documentation will be available for photocopy during site auditing and inspections, as long as subjects' names are hidden on the copy in order to maintain confidentiality.

Statistical Analysis

Analysis of Main Variable :

Acceptability Score will be summarized using a mean and a median as well as the usual indicators of variability (standard deviation, inter-quartile range, and range). The investigators will pay particular attention to the symmetry of the distribution: a strong asymmetry will suggest that the scale is not an optimal tool to measure acceptability in this sample. The analysis will be stratified in the following sub-groups: investigation site, sex, age, and duration of the disease.

Validation of the RAVIVIH Acceptability Questionnaire : Distribution of the answers, on a Likert scale, to each of the questionnaire items will be assessed through a relative frequency table in order to determine if a ceiling/flooring effect is present (i.e. more than 80% of the respondents into either extremes of the Likert scale).

Since the questionnaire is built into blocks (knowledge, perceptions, acceptability), a principal component analysis (PCA) will be performed to verify that the correlation structure of the questionnaire items' answers can allow the identification of specific dimensions. In case of strong asymmetry on the questionnaire, the analysis could be completed by a non-linear PCA. This analysis will also allow to assess the relation of questionnaire's items to acceptability and thus to justify the use of a composite score based on the answers to acceptability items. To make the interpretation of such an acceptability score easier, each score will be linearly translated to a 100-point scale.

In addition to this assessment of the RAVIVIH questionnaire's construction validity, a multitrait scaling will be performed. It will aim to verify that the correlation between items from the same dimension are appropriate (> 0.5) and that correlation between items belonging to unrelated dimensions remains low (<0.2). The statistical significance of the linear correlations will be tested with a Pearson correlation test, and correlation for multiple tests with the Bonferroni method.

Acceptability Score Validation The investigators will validate the RAVIVIH composite score (in its 100-point scale form) by comparing it with the EVA questionnaire using linear correlation coefficient (Pearson) and Spearman's rank correlation coefficient. The latter can assess the degree to which a relationship between two variables can be described by a monotonic function.

Influence of knowledge and perception of therapeutic vaccine and biomedical data on Acceptability To determine if variations in the degree of acceptability can be explained by differences in knowledge or perceptions, a canonical multivariate analysis will be performed in order to identify which items share the greatest contribution in explaining variations in the acceptability score.

Multiple correlation analyses will be performed in order to verify the association between the acceptability score and biomedical characteristics as well as quality of life as measured by the PROQOL-HIV questionnaire. Scores translating into "social relationships", "sexual relationships", "stigma", and "impact of treatment" dimensions will be of part interest. This analysis will provide, indirectly, an indication of the RAVIVIH questionnaire's convergent validity. The RAVIVIH acceptability score will also be correlated with the IPQ-R score.

Sample size assessment (total and by site) Since this study is essentially a prospective one and since it is based on a representative sample of French HIV-positive patients, the number of participants necessary was determined based on the required precision for the main indicator of therapeutic vaccine acceptability.

A sample size of 200 (N=200) allows to estimate an average acceptability score on the EVA questionnaire with a margin of error inferior to 0.5 (95% confidence interval), assuming a theoretical 1-point standard deviation. Regarding the composite acceptability score, referring to the scoring system used by Newman (2011) and assuming a standard deviation of 20 points, this translates into an average on a 100-point scale with 3-point accuracy. Furthermore, such a sample size would allow the calculation of the PCA and the extraction of 3 or 4 components.

Expected statistical significance : For all calculations and statistical tests, a 95% confidence interval will be applied.

Plan for missing data :

Missing data include variables that are reported as missing, unavailable, "non-reported", uninterpretable, or considered missing because of data inconsistency or out-of-range results. The Clinical Trial Technician or the physician will inspect the questionnaire during the consult to ensure that no items are left unanswered. If, despite this procedure, items are left unanswered, a system will be implanted so as to be able to retrieve the data necessary for statistical analysis.

Management of Modifications brought to the Initial Statistical Analysis Plan :

Modifications brought to the initial statistical analysis plan will be reported in a written document that will be attached to the initial plan. If additional statistical analysis became necessary, it would be detailed in the analysis report.

ELIGIBILITY:
Inclusion Criteria:

* infected with HIV-1
* older than 18 and younger than 75 years
* speaking , reading french
* with medical coverage (SS, CMU, AME)

Exclusion Criteria:

* protected adults (adults under guardianship, trusteeship)
* infected with HIV-2
* pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
VAS scale of acceptability | For a given participant, study procedure is about 60 minutes. Total period of the study is 12 months.
  A graduated visual analogue scale (VAS) from 0 (Whatever my situation, I never accept the use of a therapeutic vaccine) to 10 (I totally agree, and I see no problem use a therapeutic vaccine soon there will be one available).
  The VAS scale of acceptability is a classic visual analogue scale horizontal scale length 10 cm, graduated from 0 to 10, on which the patient turns his level of agreement with the proposal by a checkmark. The score can then be converted to a 100-point scale to facilitate interpretation of scores.
  Which to associate an overall acceptability score compiled from questionnaires.

SECONDARY OUTCOMES:
score of quality of life | For a given participant, study procedure is about 60 minutes. Total period of the study is 12 months.
  with the PROQOL-HIV questionnaire
confidence score of the patient-physician relationship | For a given participant, study procedure is about 60 minutes. Total period of the study is 12 months.
  with the RAVVIH questionnaire
perception score of the severity of the disease | For a given participant, study procedure is about 60 minutes. Total period of the study is 12 months.
  with the Brief IPQ-R questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: David Zucman, MD, Principal Investigator — HOPITAL FOCH Service de Medecine Interne
Locations (3):
- France (3):
  - Centre Hospitalo-Universitaire Louis Mourier, Colombes, Hauts de Seine
  - Hopital Foch, Suresnes, Hauts de Seine
  - Centre Hospitalier Regional d'Orléans, Orléans

REFERENCES:
- [Derived] Dimi S, Zucman D, Chassany O, Lalanne C, Prazuck T, Mortier E, Majerholc C, Aubin-Auger I, Verger P, Duracinsky M. Patients' high acceptability of a future therapeutic HIV vaccine in France: a French paradox? BMC Infect Dis. 2019 May 9;19(1):401. doi: 10.1186/s12879-019-4056-6. PMID 31072394